CLINICAL TRIAL: NCT03051451
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Determine the Efficacy of Two Fixed Dose Combination of Metformin/Fluoxetin 1000/40 mg vs. 1700/40 mg in the Management of Overweight and Obesity
Brief Title: Fixed Dose Combination of Fluoxetin and Metformin in the Management of Overweight and Obesity
Acronym: Metfluo
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Collaborators: INTEC Instituto de Terapéutica Experimental y Clínica, Departamento de Fisiología, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara. (Unknown); OSMO (OAXACA SITE MANAGEMENT ORGANIZATION, SC) (Unknown); IBIOMED INVESTIGACIÓN BIOMÉDICA PARA EL DESARROLLO DE FÁRMACOS, S.A. DE C.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30050/II/16
Record Dates: First submitted 2016-12-02; First posted 2017-02-13 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Overweight and Obesity
Keywords: Hydrochloride of Metformin / Fluoxetine; Placebo; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combination metformin hydrochloride/ fluoxetine 500/20 mg (Active Comparator): Dosage: The dose will depend on the period of treatment in which the patient is:
  * Single dose treatment (from visit 2 (from day 0 to day 30 ± 7), the patient will take 1 metformin hydrochloride tablet 500 mg / fluoxetine 20 mg and 1 placebo tablet , every 24 hours in the morning for 30 days).
  * Treatment at double dose (from visit 3 and until visit 8), the patient will take 2 tablets of metformin hydrochloride 500 mg / fluoxetine 20 mg and 2 tablets of Placebo, every 24 hours in the morning for 150 days).
  Interventions: Drug: combination metformin hydrochloride/ fluoxetine 500/20 mg
- combination metformin hydrochloride/ fluoxetine 1000/20mg (Active Comparator): Dosage: The dose will depend on the period of treatment in which the patient is:
  * Single dose treatment (from visit 2 (from day 0 to day 30 ± 7), the patient will take 1 metformin hydrochloride tablet 850 mg / fluoxetine 20 mg and 1 placebo tablet , every 24 hours in the morning for 30 days).
  * Treatment at double dose (from visit 3 and until visit 8), the patient will take 2 tablets of metformin hydrochloride 850 mg / fluoxetine 20 mg and 2 tablets of Placebo, every 24 hours in the morning for 150 days).
  Interventions: Drug: combination metformin hydrochloride/ fluoxetine 1000/20mg
- Placebo Oral Tablet (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: combination metformin hydrochloride/ fluoxetine 500/20 mg — Group A will receive metformin 1000 mg and 40 mg of fluoxetine; after the increment phase.
  All treatment groups will receive, in addition to the intervention, recommendations of a diet based on a hyper protein, hypo caloric and low carbohydrate diet as well as an exercise routine according to age and physical condition
  Arms: combination metformin hydrochloride/ fluoxetine 500/20 mg
Drug: combination metformin hydrochloride/ fluoxetine 1000/20mg — Group B will receive metformin 1700 mg and 40 mg of fluoxetine; after the increment phase.
  All treatment groups will receive, in addition to the intervention, recommendations of a diet based on a hyper protein, hypo caloric and low carbohydrate diet as well as an exercise routine according to age and physical condition
  Arms: combination metformin hydrochloride/ fluoxetine 1000/20mg
Drug: Placebo Oral Tablet — Group C will receive placebo oral tablet; All treatment groups will receive, in addition to the intervention, recommendations of a diet based on a hyper protein, hypo caloric and low carbohydrate diet as well as an exercise routine according to age and physical condition
  Arms: Placebo Oral Tablet

SUMMARY:
Clinical trial, multicenter, double-blind, placebo-controlled, comparative of three parallel groups, randomized treatment to assess the efficacy and safety using a fixed dose combination of metformin hydrochloride with fluoxetine as adjunctive treatment in patient with obesity or overweight in order to generate new knowledge and give a greater number of therapeutic options to the clinicians, one group will receive metformin 1700 mg and 40 mg of fluoxetine; Another group will receive metformin 1000 mg with 40 mg of fluoxetine, and a third group called control will receive placebo.

The above described treatments will be administered according to the "Dosage Schedule" The three groups will receive tablets of physical characteristics equal to the reference drug to preserve the blinding.

DETAILED DESCRIPTION:
Overweight and obesity are serious health problems that affect population around the world. According to information of the World Health Organization (WHO) in 2014 more than 1.9 billion of inhabitants older than 18 years had overweight, of which 600 million were obese, i.e., 39% of adults at global level present overweight and 13% of adults suffer obesity.

Overweight and obesity are considered complex and multifactorial diseases associated with the development of multiple co-morbidities such as certain types of cancer, cardiovascular diseases (CVD), disability, diabetes mellitus type 2 (DM2), disease of gallbladder, osteoarthritis, high blood pressure (Hypertension), sleep apnea and cerebrovascular disease (CD), making it the fifth leading cause of death worldwide , and is therefore considered a pandemic.

Obesity is defined as the increase of the weight body associated to an imbalance in the proportions of the different components of the body, in which mainly, the mass fat increases with abnormal distribution in the body.The Body Mass Index (BMI) is the standard most widely used for the classification of the somatotype in the people, and therefore the identification of obesity. BMI is obtained through by dividing the weight in kilograms between heights in squared meters. The classification of the BMI for White, Hispanic, and African-American adult people has been approved by the National Institute of Heart, Lung and Blood, the WHO, the American Association of Heart, the American College of Cardiology and the Obesity Society, whose classification is the following:

The weight body is determined by the balance energy, which represents the difference between the intake of energy through the food and the expenditure of energy coming of physical activity of an individual. For the maintenance of a stable body weight, the energy intake must be equal to energy expenditure, that's when weight gain happens, when the intake exceeds expenditure, which produces a positive energy balance. On the other hand, weight loss occurs when energy expenditure exceeds the caloric intake.

Although the low expenditure of energy represents one of the main factors that produce an increase in the weight, there are multiple factors that play an important role. These factors include genetic predisposition of the individual, physical inactivity and sedentary behavior, socio-economic factors, as well as emotional factors and consumption of certain types of drugs.

Due to the multiple factors that have an influence in the development of overweight and obesity, the treatment is complex, because there must be some type of treatment by a multidisciplinary team that achieve the control of each one of the factors that condition obesity of each individual.

Traditional treatments for loss weight have been given in the education of the individual on the preference for healthy foods, prescription diets and the implementation of programs of physical activity. However, various studies have shown that this type of intervention has few effects in long term, so the incorporation of new strategies as adjuvants in the loss of weight have been developed, which include surgical techniques and pharmacological therapies.

According to the guidelines for obesity, the drug treatment therapy should be recommended in individuals with a BMI ≥30 kg/m2 or with a BMI of ≥27 kg/m2 and the presence of a comorbidity. 6. The use of pharmacological therapies must always be used as adjuvants to changes in lifestyle, and must be approved by health authorities of each country. Before 2012, phentermine and orlistat were the unique medications available for the treatment of obesity in the United States; however in 2015 the Repertoire of pharmacological agents available to treat the obesity was extended and incorporated 4 new drugs: lorcaserin, phentermine / topiramate of prolonged release, naltrexone / wellbutrin of prolonged release and liraglutide. These new drugs share a common strategy to promote weight loss that controls hunger and satiation at the level of the central nervous system (CNS), besides that most of them have been previously used for the treatment of a medical condition other than obesity. The amount of weight lost that is achieved through the use of these agents, usually goes from 3 to 10% of the initial weight and requires a continuous to hold the loss of weight. In addition, each of these drugs has a unique profile of adverse events that should be considered deeply prior to be indicated.

Due to the above, the search for new drug therapies for the obesity treatment is one of the priorities in the research. Some drugs developed for different therapeutic indications have shown significant effects on weight loss, which include metformin hydrochloride and fluoxetine

ELIGIBILITY:
Inclusion Criteria:

* Signature of consent informed
* Men and Women.
* ≥ 18 years old proven through a current official identification.
* BMI ≥ 30 kg/m2 with or without Comorbidities.
* BMI ≥ 27 kg/m2 with a diagnosis of comorbidities by patient's clinical record associated with overweight (DM2's recent diagnosis without treatment, hypertension, dyslipidemia, sleep apnea or secondary heart disease) defined as follows:
* DM2 of current diagnosis study inclusion unless not receive drug treatment, with a HbA1c ≥6. 5 and and < 8.5%.
* Arterial Systemic Hypertension with figures < 140 / 90 mmHg.
* Dyslipidemia with total cholesterol levels> 200 mg / dl and <240 mg / dl, and / or LDL-C> 100 and <160 mg / dl and / or triglycerides> 150 mg / dl and <400 mg / dl.
* In case of have drug treatment for hypertension or dyslipidemia, the participants must have a stable dose for at least 3 months prior to the elective visit.
* Women in childbearing age must use a reliable method of birth control, such as barrier methods (condom, diaphragm), fallopian tube obstruction, intrauterine device.

Exclusion Criteria:

* Endogenous obesity (endocrine diseases that condition gain of weight, such as hypothyroidism, syndrome of Cushing).
* Background of patient's clinical record history of iatrogenic obesity (use of drugs that determine weight gain, such as corticosteroids, antipsychotic and antiepileptic).
* Thyroid stimulating Hormone (TSH) is out of range.
* Prolongation of the QT interval corrected for rate (QTc) segment by electrocardiogram with the formula of prolonged Bazett (greater than 450 msec. in males and 470 msec in women).
* Creatinine ≥1. 3 mg/dl in women and ≥1. 5 mg/dl in men.
* Alanine transaminase(ALT) or Aspartate Aminotransferase (AST) > 2 times above from the normal value.
* Background of patient's clinical record of depressive disorder or anxiety that - may require therapy with psychiatric drugs.
* Intolerance known to drugs in the study.
* Pregnancy or breastfeeding.
* Use of medications, supplements or other techniques whose objective is the reduction of weight.
* Use of medications contraindicated with drugs study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Decrease of at least 5% of body weight and the reduction in the body mass index. | six months
  Compare BMI after 6 months of treatment with hydrochloride of metformin / fluoxetine. In two doses (1000/40 mg) and (1700/40 mg) or placebo.

SECONDARY OUTCOMES:
Body weight | six months
  the mass of the body in kilograms
Height | six months
  expressed in meters
Body Mass Index | six months
  relationship between weight and height, used to classify underweight, overweight and obesity, calculated by dividing the weight in kilograms by the square of the height in meters
Waist-hip index (hip circumference) | six months
  The waist hip index will be obtained by measuring the waist perimeter in centimeters at the last floating rib level and the maximum hip perimeter at the gluteal level.
Blood pressure measurement | six months
  The blood pressure measurement will be performed with a calibrated and verified sphygmomanometer in mm/Hg
Fasting glucose concentration | six months
  Glucose concentrations in mg/dl from blood serum will be determined in patients in fasting condition
Insulin levels | six months
  Serum insulin levels in µl/ml will be quantified using an enzyme immunoassay technique
concentrations of lipid profile | six months
  Percentage of reduction of cholesterol levels in mg/dl after 6 months of treatment.
fat mass | six months
  Measured by bioimpedance
concentrations of lipid profile | six months
  Percentage of reduction LDL-C and / or triglycerides in mg/dl after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manuel González, PhD, Principal Investigator — Instituto de Terapéutica Experimental y Clínica, Departamento de Fisiología, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara.
Locations (1):
- Laboratorios SIlanes S.A. de C.V,, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Efficacy and safety using fluoxetin — http://www.medicamentosplm.com/home/productos/fluoxetina_capsulas/10/101/43902/14